CLINICAL TRIAL: NCT00361634
Title: DCE-MRI of the Wrist to Measure Short-Term Responses in Rheumatoid Arthritis Subjects Treated With Etanercept
Brief Title: Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) to Measure Response to Etanercept in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060118
Expanded Access: Available
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Etanercept; Enbrel; DCE-MRI; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (1):
- Etanercept (Experimental): Etanercept 50 mg administered by subcutaneous injection once weekly for up to 12 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept
  Other Names: Enbrel®

SUMMARY:
The purpose of this study is to assess whether DCE-MRI can detect changes of active disease in rheumatoid arthritis (RA) patients after 4, 8 and 12 weeks of etanercept.

DETAILED DESCRIPTION:
The current literature shows the promise of magnetic resonance imaging (MRI) for assessing response to therapy in RA but the heterogeneity of the methodology and the semi-quantitative nature of the image analysis limits its applicability. To evaluate the ability of DCE-MRI to serve as a biomarker for treatment-induced changes in RA associated synovial inflammation, the reproducibility of the measurement and an effect size are required. Additional endpoints such as synovial volume, bone erosion progression and bone marrow edema-like changes may also prove useful for short-term assessment of a therapeutic intervention, but have not been explored in the context of a pharmacodynamic biomarker. It is therefore critical to conduct a carefully designed longitudinal study, focused on identifying the key parameters related to the instrumentation and data analysis, to fully evaluate the potential utility of MRI in an early clinical development setting. Importantly, this study will also demonstrate the feasibility of using DCE-MRI at multiple centers to acquire useful information that will drive program decisions.

Expanded Access: Amgen provides expanded access for this clinical trial. Contact the Amgen Call Center (866-572-6436) for more information.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the 1987 American College of Rheumatology (ACR) criteria for RA with a disease duration > 6 months
* Presence of active disease (defined as both tender and swollen joints) in at least one wrist
* Sub-optimal response to methotrexate (MTX) defined by the presence of the following criteria (based on 68/66 joint count): 8 or more swollen joints AND 8 or more tender joints (with involvement of the wrist, fingers and at least one region outside the hands) at screening
* Must be receiving MTX at a stable dose > 15 mg/week at least 12 weeks prior to baseline
* a lower dose is acceptable if otherwise not tolerated (toxicity documentation required).

Exclusion Criteria:

* Patients who are currently receiving disease modifying anti-rheumatic drug (DMARD) therapy (other than MTX, hydroxychloroquine or sulfasalazine) including tumor necrosis factor (TNF) antagonists (etanercept, infliximab, and adalimumab), abatacept, rituximab, leflunomide, cyclosporine, and gold (oral and intramuscular injection) within 8 weeks or 5.5 half-lives, whichever is longer, of screening
* Co-existing condition requiring medications that alter vascular flow (e.g., nitrates, calcium channel blockers, ergot containing drugs) [Potential effects of antihypertensive and migraine medications will be discussed with the Sponsor]
* Comorbid autoimmune disorders including systemic lupus erythematosus
* Unable to undergo an MRI examination (e.g., presence of a pacemaker, defibrillator, or other implanted device such as anterior interbody cages, aneurysm clip or pedicle screws
* allergic to contrast agent
* tattoos [in area of examination if contains metallic pigment])
* or will likely require sedation for the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (2):
  - Research Site, Los Angeles, California
  - Research Site, Seattle, Washington
- Research Site, London, United Kingdom

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 13 December 2006 through 27 April 2009
Period: Overall Study
Arm/Group | Etanercept
Started | 14
Treated | 13 (The safety analysis set consisted of all patients who received at least one dose of etanercept.)
Completed | 12
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 8
  Black or African American | 1
  Hispanic or Latino | 4
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Synovial Transfer Constant (Ktrans) From Days 1-29
Description: Percent change in transfer constant (Ktrans) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from study day 1 to study day 29. Ktrans reflects contrast delivery (capillary blood flow) and transport across the vascular endothelium (capillary permeability-surface area product), with the dominant factor depending on whether delivery is flow or permeability limited. A Ktrans value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, an increase in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Day 1 to Day 29
Population: Full Analysis Set, composed of all participants who had a baseline and at least one post-baseline measurement. Only participants with available Day 29 data are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percent change | 15.04 (70.53)

2. Secondary Outcome: Percent Change in Synovial Volume From Days 1-29
Description: Percent change in the synovial volume for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from Day 1 to Day 29. Synovial volume was evaluated by image subtraction from the T1-weighted images pre-and post-administration of the contrast agent.
Time Frame: Day 1 to Day 29
Population: Full Analysis Set, composed of all participants who had a baseline and at least one post-baseline measurement. Only participants with available data are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percent change | -4.15 (46.54)

3. Primary Outcome: Percent Change in Synovial Transfer Constant (Ktrans) From Days 1-57
Description: Percent change in transfer constant (Ktrans) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from study day 1 to study day 57. Ktrans reflects contrast delivery (capillary blood flow) and transport across the vascular endothelium (capillary permeability-surface area product), with the dominant factor depending on whether delivery is flow or permeability limited. A Ktrans value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, an increase in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Day 1 to Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Percent change | 40.75 (77.28)

4. Primary Outcome: Percent Change in Synovial Transfer Constant (Ktrans) From Days 1-85
Description: Percent change in transfer constant (Ktrans) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from study day 1 to study day 85. Ktrans reflects contrast delivery (capillary blood flow) and transport across the vascular endothelium (capillary permeability-surface area product), with the dominant factor depending on whether delivery is flow or permeability limited. A Ktrans value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, increases in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Percent change | 55.00 (136.97)

5. Primary Outcome: Percent Change in Synovial Initial Area Under the (Contrast-time) Curve (IAUC) From Days 1-29
Description: Percent change in the synovial initial area under the contrast-time curve (IAUC) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from Day 1 to Day 29. IAUC reflects the contrast distribution volume (extravascular extracellular space) in addition to contrast delivery and transport across the vascular endothelium. An IAUC value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, an increase in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Day 1 to Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 13
Percent change | 8.64 (59.65)

6. Primary Outcome: Percent Change in the Synovial Initial Area Under the Contrast-Tme Curve (IAUC) From Days 1-57
Description: Percent change in the synovial initial area under the contrast-time curve (IAUC) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from Day 1 to Day 57. IAUC reflects the contrast distribution volume (extravascular extracellular space) in addition to contrast delivery and transport across the vascular endothelium. An IAUC value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, an increase in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Day 1 to Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Percent change | 15.30 (33.98)

7. Primary Outcome: Percent Change in the Synovial Initial Area Under the Contrast-Time Curve (IAUC) From Days 1-85
Description: Percent change in the synovial initial area under the contrast-time curve (IAUC) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from Day 1 to Day 85. IAUC reflects the contrast distribution volume (extravascular extracellular space) in addition to contrast delivery and transport across the vascular endothelium. An IAUC value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, an increase in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Percent change | 34.54 (84.91)

8. Secondary Outcome: Percent Change in Synovial Volume From Days 1-57
Description: Percent change in the synovial volume for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from Day 1 to Day 57. Synovial volume was evaluated by image subtraction from the T1-weighted images pre-and post-administration of the contrast agent.
Time Frame: Day 1 to Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 11
Percent change | -6.52 (31.47)

9. Secondary Outcome: Percent Change in Synovial Volume From Days 1-85
Description: Percent change in the synovial volume for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) of the wrist from Day 1 to Day 85. Synovial volume was evaluated by image subtraction from the T1-weighted images pre-and post-administration of the contrast agent.
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
Percent change | 7.75 (55.33)

10. Secondary Outcome: Difference Between Percent Change in Ktrans From Days -28 to 1 and Days 1 to 29
Description: Difference in percent change between synovial transfer constant (Ktrans) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from study day 1 to study day 29 and from study day -28 to study day 1.
Time Frame: Day -28 to Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 13
percent change | -50.24 (231.80)

11. Secondary Outcome: Difference Between Percent Change in Ktrans From Days -28 to 1 and Days 1 to 57
Description: Difference in percent change between synovial transfer constant (Ktrans) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from study day 1 to study day 57 and from study day -28 to study day 1.
Time Frame: Day -28 to Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
percent change | -49.96 (265.51)

12. Secondary Outcome: Difference Between Percent Change in Ktrans From Days -28 to 1 and Days 1 to 85
Description: Difference in percent change between synovial transfer constant (Ktrans) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from study day 1 to study day 85 and from study day -28 to study day 1
Time Frame: Day -28 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
percent change | -35.72 (293.47)

13. Secondary Outcome: Difference Between Percent Change in IAUC From Days -28 to 1 and Days 1 to 29
Description: Difference in percent change between the synovial initial area under the contrast-time curve (IAUC) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from Day 1 to Day 29 and from Day -28 to Day 1
Time Frame: Day -28 to Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 13
percent change | -5.96 (126.57)

14. Secondary Outcome: Difference Between Percent Change in IAUC From Days -28 to 1 and Days 1 to 57
Description: Difference in percent change between the synovial initial area under the contrast-time curve (IAUC) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from Day 1 to Day 57 and from Day -28 to Day 1
Time Frame: Day -28 to Day 57
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
percent change | -8.68 (127.57)

15. Secondary Outcome: Difference Between Percent Change in IAUC From Days -28 to 1 and Days 1 to 85
Description: Difference in percent change between the synovial initial area under the contrast-time curve (IAUC) for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from Day 1 to Day 85 and from Day -28 to Day 1
Time Frame: Day -28 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 10
percent change | 10.55 (146.25)

ADVERSE EVENTS:
Time Frame: From first dose date to 30 days after last dose (up to 16 weeks).
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 12/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=13)
Palpitations (Cardiac disorders) | 1
Myodesopsia (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 2
Injection site haematoma (General disorders) | 1
Injection site reaction (General disorders) | 3
Injection site urticaria (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Breast tenderness (Reproductive system and breast disorders) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial resul